CLINICAL TRIAL: NCT02343419
Title: Diagnostic Utility of Different Airway Resistance Assessment Techniques in the Evaluation of Bronchial Hyperreactivity by Methacholine Challenge Testing
Brief Title: Diagnostic Utility of Different Airway Resistance Assessment Techniques in the Methacholine Challenge Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PFT-DIMPA-WUM1
Record Dates: First submitted 2014-12-01; First posted 2015-01-22 (Estimated); Last update posted 2016-11-09 (Estimated); Status verified 2016-11

CONDITIONS: Bronchial Hyperreactivity; Abnormal Respiratory Airway Resistance
Keywords: Bronchial Hyperreactivity; Bronchial Provocation Tests; Methacholine Chloride; Respiratory Function Tests; Spirometry; Airway Resistance; Plethysmography
MeSH Terms: conditions — Bronchial Hyperreactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bronchial challenge test (Experimental): Patients will undergo Methacholine Challenge Test assessed by forced oscillation technique (FOT), plethysmography, interrupter technique and spirometry.
  Interventions: Other: Methacholine Challenge Test

INTERVENTIONS:
Other: Methacholine Challenge Test — Forced oscillation technique test, plethysmography, interrupter technique test and spirometry will be performed in a row before any intervention and after inhalation of aerosols - normal saline, followed by increasing concentrations of methacholine: 0.03 mg/ml; 0.06 mg/ml; 0.125 mg/ml; 0.25 mg/ml, 0.5 mg/ml, 1 mg/ml, 2 mg/ml, 4 mg/ml, 8 mg/ml, 16 mg/ml.
  In case of FEV1 decrease of ≥ 20% of the initial value methacholine challenge test will be ceased and patient will be administered 200 µg of salbutamol in inhalation. Then, pulmonary function tests will be performed after 15 minutes.

SUMMARY:
The aim of the study is to compare standard spirometric evaluation of methacholine challenge test with plethysmographic, interrupter technique and forced oscillation technique (FOT) evaluation of the airways resistance.

The study group will consist of patients referred for methacholine challenge test. All patient will undergo spirometric, plethysmographic, interrupter technique and FOT examinations - before and after inhalation of aerosols. Patients will also undergo the measurement of nitric oxide concentration in exhaled air and laboratory tests, including: blood count, measurement of serum C-reactive protein, sodium, potassium, creatinine, immunoglobulin E and N-Terminal pro-brain natriuretic peptide (NT-proBNP) concentration.

The investigators intend to assess, if plethysmographic, and/or interrupter, and/or FOT measurement of bronchial reactivity can replace standard spirometric assessment. Plethysmography, interrupter technique and FOT are much more easier to perform for patients. Furthermore, those two techniques are less dependent on patient's motivation and cooperation ability. Thus, usage of FOT, interrupter technique and/or plethysmography in bronchial hyperreactivity testing could make methacholine challenge test more comfortable and available for more patients. The investigators are also going to analyze the relationship between exhaled nitric oxide and functional indices of bronchial hyperreactivity.

DETAILED DESCRIPTION:
Bronchial hyperreactivity is defined as the increased respiratory tract responsiveness to multiple stimuli, which results in bronchial muscles constriction and bronchial lumen narrowing. Bronchial hyperreactivity is a hallmark of asthma, however it may also be present in other diseases, e.g. chronic obstructive pulmonary disease (COPD). Methacholine challenge test is one of the bronchial reactivity assessment methods. Methacholine acts directly on bronchial smooth muscles receptors and causes bronchoconstriction. Bronchial reactivity is increased in the presence of active inflammation. Methacholine challenge testing is commonly performed in patients with symptoms suggestive of asthma and negative result of spirometry reversibility test. The measurement of methacholine concentration which causes 20% forced expiratory volume at one second (FEV1) decrease in post-inhalation spirometry (PC20) is a standard method of hyperreactivity evaluation. However, above method could be used among patients who are able to perform acceptable spirometry. Furthermore, results of spirometry might be influenced by level of compliance and motivation of patients. Moreover, whereas spirometric methacholine challenge test has high negative predictive values, its positive predictive value is relatively low. Thus, diagnostic utility of other pulmonary function tests should be assessed in methacholine challenge test evaluation.

In plethysmography airway resistance is performed during tidal breathing. The increase of specific airway resistance of 200% and the decrease of specific airway conductance of 40% after methacholine inhalation, respectively, are proposed as a cut-off levels for bronchial hyperreactivity diagnosis.

In forced oscillation technique (FOT), sinusoidal oscillations are emitted by membrane into airway lumen and airway resistance is calculated on the basis of changes in air flow induced by oscillations. The increase of resistance and decrease of reactance in FOT are typical for bronchoconstriction.

Finally, also interrupter technique (IT) allows for airway resistance assessment during tidal breathing. In IT, airway resistance is calculated on the basis of mouth pressure measured directly after airway occlusion and airflow measured directly before occlusion.

The aim of the study is to compare standard spirometric evaluation of methacholine challenge test with plethysmographic, interrupter technique and forced oscillation technique (FOT) evaluation of the airways resistance.

All patient will undergo:

* clinical examination
* measurement of nitric oxide concentration in exhaled air
* spirometric, plethysmographic, interrupter technique and FOT examinations - before inhalation and after inhalation of aerosols
* following laboratory tests: blood count, measurement of serum C-reactive protein (CRP), sodium, potassium, creatinine, immunoglobulin E and NT-proBNP concentration

Patients will be provided with written and spoken information about study protocol. Written informed consent will be obtained from every patient.

ELIGIBILITY:
Inclusion Criteria:

* presence of asthma symptoms without confirmation of diagnosis by standard methods
* dyspnea and/or cough of unknown etiology

Exclusion Criteria:

* FEV1 <1.2 L or <60% of predicted value
* acute heart failure
* myocardial infarction in last 3 months
* transient ischaemic attack or stroke in last 3 months
* aneurysms
* methacholine allergy
* pregnant and lactating women
* administration of β2-mimetic, anticholinergic agent or theophylline before methacholine challenge test in 6, 8 and 24 hours, respectively
* respiratory tract infection in last 6 weeks
* patient inability to cooperate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2014-11; Primary Completion 2016-01 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
The concentration of methacholine inducing a 20% fall in FEV(1) from post-diluent baseline [PC(20)] | up to 2 hours
  In case of FEV1 decrease of > 20% from baseline PC (20) will be calculated by logarithmic interpolation.

SECONDARY OUTCOMES:
Change in FOT resistance and reactance from post-diluent baseline after inhalating consecutive methacholine aerosols | within 6 minutes after methacholine aerosol inhalation
  Airway resistance and reactance will be measured by FOT after inhalating methacholine aerosols until FEV(1) fall of >20% from baseline
Change in plethysmographic airway resistance from post-diluent baseline after inhalating consecutive methacholine aerosols | within 6 minutes after methacholine aerosol inhalation
  Airway resistance will be measured by plethysmography after inhalating methacholine aerosols until FEV(1) fall of >20% from baseline
Change in interrupter airway resistance from post-diluent baseline after inhalating consecutive methacholine aerosols | within 6 minutes after methacholine aerosol inhalation
  Airway resistance will be measured by interrupter technique after inhalating methacholine aerosols until FEV(1) fall of >20% from baseline
Change in FEV(1) from from post-diluent baseline after inhalating consecutive methacholine aerosols | within 6 minutes after methacholine aerosol inhalation
  FEV (1) will be measured by spirometry after inhalating methacholine aerosols until FEV(1) fall of >20% from baseline
Assessment of the difficulty level of FOT | after methacholine challenge test (up to 2 hours two hours from the start of the methacholine challenge test)
  Patients will receive visual analogue scale form assessing difficulty level and problems related to performing each test
Assessment of the difficulty level of plethysmography | after methacholine challenge test (up to 2 hours two hours from the start of the methacholine challenge test)
  Patients will receive visual analogue scale form assessing difficulty level and problems related to performing each test
Assessment of the difficulty level of interrupter technique | after methacholine challenge test (up to 2 hours two hours from the start of the methacholine challenge test)
  Patients will receive visual analogue scale form assessing difficulty level and problems related to performing each test
Assessment of the difficulty level of spirometry | after methacholine challenge test (up to 2 hours two hours from the start of the methacholine challenge test)
  Patients will receive visual analogue scale form assessing difficulty level and problems related to performing each test
Duration of the bronchial resistance assessment by FOT | During methacholine challenge test (up to 2 hours)
  Duration of each pulmonary function test will be measured
Duration of the bronchial resistance assessment by plethysmography | During methacholine challenge test (up to 2 hours)
  Duration of each pulmonary function test will be measured
Duration of the bronchial resistance assessment by interrupter technique | During methacholine challenge test (up to 2 hours)
  Duration of each pulmonary function test will be measured
Duration of spirometry | During methacholine challenge test (up to 2 hours)
  Duration of each pulmonary function test will be measured
Total duration of methacholine challenge test | During methacholine challenge test (up to 2 hours)
  Total duration bronchial challenge will be measured

OTHER OUTCOMES:
Measurement of nitric oxide concentration in exhaled air | Participanst will undergo measurement of nitric oxide concentration in exhaled air immediately before bronchial challenge test, total time of measurement: approximately 10 minutes
  Nitric oxide concentration in exhaled air will be measured once, immediately before performing methacholine challenge test
Laboratory tests | Patients will undergo laboratory tests once before perfoming methacholine challenge test; maximum period between the methacholine challenge test and performing laboratory tests: one month
  Following laboratory tests will be performed: blood count, measurement of serum C-reactive protein, sodium, potassium, creatinine, immunoglobulin E and NT-proBNP concentration

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz A Urbankowski, MD, Principal Investigator — Department of Internal Medicine, Pneumonology and Allergy, Medical University of Warsaw
Locations (1):
- Department of Internal Medicine, Pneumonology and Allergy, Medical University of Warsaw, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Urbankowski T, Przybylowski T. Methacholine Challenge Testing: Comparison of FEV1 and Airway Resistance Parameters. Respir Care. 2021 Mar;66(3):449-459. doi: 10.4187/respcare.08331. Epub 2020 Nov 17. PMID 33203723